CLINICAL TRIAL: NCT00192881
Title: Stenting With or Without Coating Compared With Angioplasty in Non-benestent Disease. A Randomised Comparison of Optimal Balloon Angioplasty and Primary Implantation of Stents With and Without Drug Elution in Complex Coronary Lesions
Brief Title: Stenting With or Without Coating Compared With Angioplasty in Non-benestent Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCANDSTENT A
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2010-08-18 (Estimated); Status verified 2010-07

CONDITIONS: Coronary Artery Disease
Keywords: Percutaneous coronary intervention; Balloon angioplasty; Restenosis; Stents
MeSH Terms: conditions — Coronary Artery Disease

INTERVENTIONS:
Device: Bx Sonic & Cypher stent from Cordis

SUMMARY:
The purpose of this study is to evaluate the clinical and angiographic outcome of implantation of stents eluting or not eluting Sirolimus in patients with complex coronary artery lesions suitable for percutaneous coronary intervention.

ELIGIBILITY:
Inclusion Criteria:

* Stable, or unstable angina and/or objective signs of myocardial ischaemia
* Informed consent
* Optimal result (< 35% residual stenosis and < type C dissection) after balloon angioplasty
* Lesions should be de novo and located in native vessels with a diameter > 2.25 mm.
* Complex lesions to be included should have at least one of the following characteristics:

  * ostial in location (< 5 mm from ostium)
  * total occlusions with a length ≥ 15 mm
  * bifurcational (side branch > 1.75 mm in diameter)
  * angulated (> 45° within lesion)

Exclusion criteria:

Patients:

* Other severe disease with an expected survival < 1 year
* Other significant cardiac disease
* Known allergy against paclitaxel, clopidogrel (or ticlopidine),
* Myocardial infarction within 3 days of the index procedure
* Linguistic difficulties needing an interpreter
* Renal insufficiency (p-creatinine > 200 micromol/l)
* Gastrointestinal bleeding within 1 month
* Childbearing potential or pregnancy
* Participation in another study

Lesions:

* Unprotected left main disease
* Restenosis
* Lesions containing visible thrombus
* Treatment with other modality than balloon or stent (ablation, brachytherapy, ultrasound) in connection with the index procedure
* Diffuse coronary disease distal to the treated lesion
* Heavily calcification
* Lesion located in saphenous vein graft

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-10

CONTACTS AND LOCATIONS:
Overall Officials: Henning Kelbaek, MD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Cardiac Cath Lab, Copenhagen, Denmark